CLINICAL TRIAL: NCT00153660
Title: A Double-blind Randomized Comparison of Celecoxib Plus Esomeprazole Versus Naproxen Plus Esomeprazole for Prevention of Recurrent Ulcer Bleeding in Patients With Arthritis and Cardiothrombotic Diseases (NSAID#8 Study)
Brief Title: Celecoxib Versus Naproxen for Prevention of Recurrent Ulcer Bleeding in Arthritis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Francis KL Chan, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8N Study
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Arthritis; Cardiovascular Diseases; Cerebrovascular Disorders
MeSH Terms: conditions — Arthritis; Cardiovascular Diseases; Cerebrovascular Disorders | interventions — Celecoxib; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NSAID #1 (Active Comparator): Celecoxib and Naproxen Placebo
  Interventions: Drug: Celecoxib(drug)
- NSAID #2 (Active Comparator): Naproxen and Celecoxib Placebo
  Interventions: Drug: Naproxen(drug)

INTERVENTIONS:
Drug: Celecoxib(drug) — Celecoxib 100 mg bd
  Other Names: Celebrex
  Arms: NSAID #1
Drug: Naproxen(drug) — Naproxen 500 mg bd
  Other Names: Naprosyn
  Arms: NSAID #2

SUMMARY:
The aim of this study is to compare celecoxib plus a PPI (esomeprazole) versus naproxen plus a PPI (esomeprazole) in preventing recurrent ulcer bleeding in arthritis patients with a history of ulcer bleeding who require concomitant ASA. We hypothesized that among patients with a history of ulcer bleeding who require concomitant ASA, celecoxib plus esomprazole would be superior to naproxen plus esomeprazole for the prevention of recurrent ulcer bleeding.

DETAILED DESCRIPTION:
Nonsteroidal anti-inflammatory drugs (NSAIDs) are the most commonly consumed drugs worldwide for the relief of pain and arthritis. However, the use of NSAIDs increases the risk of ulcer bleeding by 4-fold. Current evidence indicates that combination of conventional NSAIDs and a proton pump inhibitor (PPI) reduces the risk of ulcer complications. The alternative strategy is to replace conventional, non-selective NSAIDs with NSAIDs selective for cyclooxygenase-2 (COX-2 inhibitors). Recently, there are concerns about the cardiovascular safety of COX-2 inhibitors and conventional NSAIDs. Because of such concern, patients requiring anti-inflammatory analgesics who have cardiovascular risk factors (e.g. smoking, hypertension, hyperlipidemia, diabetes) should receive prophylactic low-dose aspirin. However, concomitant low-dose aspirin negates the gastric sparing effect of COX-2 inhibitors and augments the gastric toxicity of nonselective NSAIDs. Thus, gastroprotective agents such as PPIs should be co-prescribed to patients with high ulcer risk who are taking aspirin plus a COX-2 inhibitor or a nonselective NSAID.

ELIGIBILITY:
Inclusion Criteria:

1. age >18,
2. a history of endoscopically proven gastroduodenal ulcer bleeding,
3. H. pylori negative
4. a history of cardiothrombotic disease requiring ASA, and
5. anticipated regular use of NSAIDs for the duration of trial

Exclusion Criteria:

1. concomitant use of anticoagulants;
2. a history of gastric or duodenal surgery other than a patch repair;
3. the presence of erosive esophagitis,
4. gastric outlet obstruction,
5. renal failure (defined by a serum creatinine level of more than 200 umol/L),
6. pregnancy,
7. terminal illness, or
8. cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2005-06; Primary Completion 2014-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Recurrent ulcer bleeding within 18 months according to pre-specified criteria | 18 months

SECONDARY OUTCOMES:
patients' global assessment of arthritis | 18 months
major CV events according to the Antithrombotic Trialists' criteria | 18 months
non-fatal myocardial infarction | 18 months
non-fatal stroke | 18 months
death from a vascular cause | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Francis K Chan, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Center, Prince of Wales Hospital, Shatin, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan FKL, Ching JYL, Tse YK, Lam K, Wong GLH, Ng SC, Lee V, Au KWL, Cheong PK, Suen BY, Chan H, Kee KM, Lo A, Wong VWS, Wu JCY, Kyaw MH. Gastrointestinal safety of celecoxib versus naproxen in patients with cardiothrombotic diseases and arthritis after upper gastrointestinal bleeding (CONCERN): an industry-independent, double-blind, double-dummy, randomised trial. Lancet. 2017 Jun 17;389(10087):2375-2382. doi: 10.1016/S0140-6736(17)30981-9. Epub 2017 Apr 11. PMID 28410791